CLINICAL TRIAL: NCT06279624
Title: Effectiveness of the 13-Valent Pneumococcal Conjugated Vaccine Against Community-Acquired Pneumonia in Older Thai Adults: A Matched Case-Control Study.
Brief Title: Effectiveness of the PCV13 in Older Thai Adults
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Sponsor
Other Study IDs: NRCT9-4
Record Dates: First submitted 2024-01-05; First posted 2024-02-28 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is the matched 1:2 case-control study, prospectively collect case and control who are diagnosed with pneumococcal or non-pneumococcal community acquired pneumonia (CAP), accordingly from November 2023 through October 2024. The investigators define a CASE as a person aged ≥60 years due to pneumococcal confirmed CAP either in-patients or out-patients by doctor in charge. While a CONTROL is defined as a person aged ≥60 years due to non-pneumococcal confirmed CAP either in-patients or out-patients by doctor in charge.

The goal of this observational study is to evaluate the effectiveness of the 13-valent pneumococcal conjugate vaccine (PCV13) in pneumococcal CAP in Thai adults aged ≥ 60 years with or without any medical conditions.

The main questions it aims to answer is:

• What are the effectiveness of PCV13 for preventing all typed, vaccine typed, or non-vaccine typed of pneumococcal CAP among Thai older adults?

The investigators retrospectively collect cases and control who are diagnosed with CAP accordingly from January 2012 through October 2023. The investigators define case and control the same as prospective method, but all data were retrieved from archive database.

-The investigators select a 1:2 matched control with criteria as follows; 10-year-interval of age, ward (the same patient care such as out or in-patient, or admitted in the same level ward).

Participants will be

* collated from hospital database regarding their CAP illnesses by pneumococcal and non-pneumococcal pneumonia condition.
* explored their vaccine status by either vaccine book checking or hospital database.

Researcher will compare the effectiveness of PCV13 to prevent all typed, vaccine typed and non-vaccine typed pneumococcal pneumonia.

DETAILED DESCRIPTION:
The investigators select a 1:2 matched control with criteria as follows; 10-year-interval of age, ward (the same patient care such as out or in-patient, or admitted in the same level ward).

Patient data will be collected through review of medical records and interview of the patients or their relatives for visits to the doctors using standard Case Record Form (CRF) by trained research assistance.

Definition of CAP is defined according to clinical evidence and radiological evidence17. The clinical evidence consists of ≥2 of the following: fever, hypothermia, chills or rigors, pleuritic chest pain, cough, sputum production, dyspnea, tachypnea, malaise, or abnormal auscultatory findings suggestive of pneumonia; while the radiological evidence includes a chest radiograph and/or a computed tomographic image with an infiltrate consistent with pneumonia as determined by the treating healthcare provider or radiologist at the time of presentation. The investigators consider PCV13 status when the vaccine has been given ≥14 days before onset of CAP for cases or ≥14 days before the date of admission for control. The PCV13 status is ascertained by staff blinded to whether the patients are case or control. Status will be confirmed by hospital record or vaccination card. If history of vaccination is verbal confirmation by patient or their relatives, then the investigators plan to figure vaccine status out in all hospitals that individuals has visited before admission.

ELIGIBILITY:
Inclusion Criteria:

Prospective collection For case

1. Thai older adults aged ≥60 years with or without health conditions diagnosed with culture confirmed pneumococcal community acquired pneumonia during 2012 - 2024.
2. Be given treatment either in-hospital admission or out-patient visiting hospital.
3. They ensure their PCV13 status (either received or not received is acceptable)
4. Willing to participate in the study by their own decision or as a legal guardian.

For matched control

1. Thai older adults aged ≥60 years with or without health conditions diagnosed with non-pneumococcal community acquired pneumonia by doctor in-charge during 2012 - 2024.
2. Be given treatment either in-hospital admission or out-patient visiting in the same hospital with matched-case.
3. They ensure their PCV13 status (either received or not received is acceptable)
4. Willing to participate in the study by their own decision or as a legal guardian.

Retrospective collection For case

1. Thai older adults aged ≥60 years with or without health conditions diagnosed with culture confirmed pneumococcal community acquired pneumonia during 2012 - 2024.
2. Be given treatment either in-hospital admission or out-patient visiting hospital.
3. Certain documented PCV13 status (either received or not received is acceptable)
4. Recorded ICD: J13

For matched control

1. Thai older adults aged ≥60 years with or without health conditions diagnosed with non-pneumococcal community acquired pneumonia by doctor in-charge during 2012 - 2024.
2. Be given treatment either in-hospital admission or out-patient visiting in the same hospital with matched-case.
3. Certain documented PCV13 status (either received or not received is acceptable)
4. Recorded ICD: J09-18 (except J13)

Exclusion Criteria:

For case

1. Unknown PCV13 status/history
2. Timing between PCV13 and the onset of community acquired pneumonia <14 days.
3. Unable to collect confirmed pneumococcal samples from microbiology laboratory.

For control

1. Unknown PCV13 status/history
2. Timing between PCV13 and the onset of community acquired pneumonia <14 days.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Thai older adults aged ≥60 years with or without health conditions
  2. Diagnosed with all caused community acquired pneumonia by doctor in-charge.
  3. Either in-hospital admission or out-patient care
  4. Confirmed PCV13 vaccine history documented by verbal or vaccination record.
Sampling Method: Non-Probability Sample
Enrollment: 825 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Vaccine effectiveness of PCV13 on all types of pneumococcal CAP | April - June 2025
  All types of pneumococcal CAP will be determined by the total number of confirmed pneumococcal CAP cases regardless of serotypes over study period (unit: number of cases). Then, CAP cases will be stratified by history of vaccine. Vaccine effectiveness (VE) is calculated as follows; VE = 1- OR. OR (odds ratio) define as pneumococcal confirmed CAP among PCV13 vaccinated group/ pneumococcal confirmed CAP among without PCV13 vaccinated group.

SECONDARY OUTCOMES:
Vaccine effectiveness of PCV13 on PCV13 (vaccine typed) and non-PCV13 (non-vaccine typed) pneumococcal CAP | April - June 2025
  Vaccine types of pneumococcal CAP will be measured by the number of confirmed pneumococcal CAP cases in which pneumococcal serotype identified in vaccine (PCV13) over study period (unit: number of cases). Non-vaccine types of pneumococcal CAP will be measured by the number of confirmed pneumococcal diagnosed CAP cases in which pneumococcal serotype unidentified in vaccine (PCV13) over study period (unit: number of cases). Vaccine effectiveness will be calculated the same way as primary outcome measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, Prof., Study Chair — Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University
Locations (1):
- Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided